CLINICAL TRIAL: NCT05683314
Title: A Comparison Study for Unstable Sacrum/Pelvis and Acetabular Fracture Treated With Open Reduction and Internal Fixation With Minimally Invasive Internal Fixation
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chun-Hao Tsai, Medical doctors, Department of Orthopedics , Principal Investigator, Clinical Professor, China Medical University Hospital
Other Study IDs: CMUH108-REC3-144
Record Dates: First submitted 2022-12-23; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Unstable Sacral/Pelvic or Acetabular Fracture
Keywords: Unstable sacral; Unstable pelvic; acetabular fracture
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acetabular_Pelvic_Sacral fracture with open reduction and internal fixation
  Interventions: Procedure: Tranditional open reduction and internal fixation
- Acetabular_Pelvic_Sacral fracture with minimally invasive internal fixation

INTERVENTIONS:
Procedure: Tranditional open reduction and internal fixation — Under navigation and bone desity projecting method assisted 3D simulation and printing for minimal invasive surgrey
  Other Names: Minimally invassive internal fixation; Navigation; 3D printing modle; 3D simulation
  Groups: Acetabular_Pelvic_Sacral fracture with open reduction and internal fixation

SUMMARY:
Unstable sacral/pelvic or acetabular fracture are severe high energy fractures Surgical intervention are necessary after patient's conditions are stable. The complexity of local anatomical structure, the nearby major vessels, organ and visceral structures make the operations difficult and in high risks.

DETAILED DESCRIPTION:
The surgical principles are concluded as:

1. Sacrum fracture with rotational instability: close reduction and iliosacral screw fixation
2. Sacrum fracture with vertical shearing instability: open reduction and ipsilateral riangular osteosynthesis with /without neurological decompression
3. Spinopelvic dissociation: open reduction and bilateral triangular osteosynthesis with

   /without neurological decompression
4. Iliac fracture with sacroiliac joint(SI) joint dislocation: close reduction with iliosacral screw fixation (for SI joint dislocation), anterior open reduction with double plates fixation (for iliac fracture)
5. Anterior acetabular/ pubic fracture: close /open reduction with plates/screw fixation.
6. Symphysis dislocation: open reduction with double plates
7. Acetabulum fracture: posterior open reduction with double plates anterior open /minimally invasive reduction with plates/screw fixation. The implementation of anterior column screw under C-arm X-ray transillumination for pubic fractures was first report in the literature in 1995, and we had this surgical method in our hospital since 2011. The first report of minimally invasive internal fixation in pelvic or acetabular in the literature was reported in 2013, and we had such minimally invasive surgical approach in our hospital since 2014. We would like to retrospectively and prospectively collect the final outcome of these patients and the comparative analysis of different surgical methods in our institution.

AO foundation published an updated fracture and dislocation classification compendium in 2018. Pelvic ring fracture is classified into ABC three type according to intact, incomplete/complete disruption of the posterior arch. Each type of injury is further divided into groups regarding of severity. The old Young Burgess classification of pelvic ring injury has been integrated into this classification. This retrospective study aim to re-classify patients who sustained unstable pelvic fracture and underwent surgery in CMUH under Dr. Tsai since 2009 according to the new system.

The investigators adopted Majeed Pelvic Score for functional outcome and EQ-5D for quality of life evaluation. A telephone survey will be conducted for all patients. Multiple logistic and linear regression analyses will be used for statistical assessment with the MPS and the EQ-5D. This will provide the investigators with the insight of the correlation between injury severity and functional/QOL outcome. Also, the investigators' study aims to determine the prognostic factors relate to poor outcome. Age, mechanism of injury, sex, ISS score, associated injury, surgical method, bladder or neurologic complication, radiologic outcome,unity of fracture will be recorded from medical chart. Statistical analysis will be conducted to identify the correlation between each factor that influence the functional and QOL outcome.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above with the appropriate informed consent
2. traumatic pelvic or acetabular fracture with 2018 AO/OTA classification
3. a minimum of 48 months postoperative follow-ups

Exclusion Criteria:

1. pelvic or acetabular fractures that were pathological or non-traumatic in nature
2. patients with incomplete follow-up details
3. patients who denied surgical management
4. patients who received external fixation as part of their treatment strategy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sacral/pelvic or acetabular fracture patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
EQ-VAS | Post-operative at 48th month
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
EQ-5D | Post-operative at 48th month
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used.
Majeed pelvic score | Post-operative at 48th month
  he Majeed scoring system is a disease-specific outcome measure that was originally designed to assess pelvic injuries.

SECONDARY OUTCOMES:
Blood loss | intraoperative blood loss
  We used a cut-off of 500 cc blood loss. 500 cc was determined in accordance to the American College of Surgeons Advanced Trauma Life Support haemorrhagic shock classification, whereby a 10 to 15% blood volume loss of 500 to 750 cc in a healthy 70 KG human adult would lead to physiological changes.
Surgical duration | intraoperative duration
  4 hours of surgical duration was determined according to a review by Cheng et al. in which 2 to 4 hours of surgery was shown to lead to increased risks of postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: No